CLINICAL TRIAL: NCT06074120
Title: Assessing the Efficacy of Low-Level Laser Therapy in Alleviating Genitourinary Symptoms of Menopause
Brief Title: Low-level Laser Therapy in Genitourinary Symptoms of Menopause
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Beihu Branch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202307193DIND
Record Dates: First submitted 2023-09-24; First posted 2023-10-10 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Menopause Related Conditions
Keywords: Genitourinary symptom; Vulvovaginal atrophy; Menopause
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with genitourinary symptoms of menopause (Experimental): Receive low-level laser therapy
  Interventions: Device: Low-level laser therapy

INTERVENTIONS:
Device: Low-level laser therapy — Low-level laser therapy would be introduced via a vaginal probe (gain medium: Gallium-Aluminum-Arsenide, wavelength 660nm) for 30 minutes per treatment, once a week, for 8 courses.

SUMMARY:
The study will employ a prospective single-arm design involving menopausal women who present with genitourinary symptoms of menopause (GSM). Due to the preliminary nature of this study and the absence of a control group, the primary objective is to evaluate the feasibility and potential efficacy of low-level laser therapy in alleviating GSM in this population.

DETAILED DESCRIPTION:
A convenience sample of menopausal women aged more or equal to 45 years will be recruited from the gynecology clinic in our hospital and its branches. Participants will undergo an initial screening to confirm the presence of genitourinary symptoms associated with menopause. Inclusion criteria will encompass women experiencing symptoms such as urinary incontinence, vaginal dryness, dyspareunia, and decreased sexual satisfaction. The exclusion criteria will be diagnosed with advanced pelvic organ prolapse (more or equal to stage 2 prolapse by pelvic organ prolapse quantification system).

All participants will receive low-level laser therapy (LLLT) as the intervention. LLLT sessions will be conducted once a week for eight weeks. The laser therapy will be administered by a trained healthcare professional using a standard protocol, targeting the genitourinary area. The laser device will emit low-energy laser light, which is hypothesized to stimulate tissue regeneration, improve blood circulation, and alleviate symptoms in the genitourinary region.

Baseline assessments will be conducted prior to the initiation of LLLT, including demographic data collection and validated outcome measures to evaluate GSM and quality of life. These measures may include the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF), Female Sexual Function Index (FSFI), Vaginal Health Index (VHI), Incontinence Impact Questionnaire-7 (IIQ-7), Overactive Bladder Symptom Score (OABSS), Urogenital Distress Inventory-6 (UDI-6), Urgency Severity Scale (USS), King's Health Questionnaire (KHQ), and a urodynamic study with a 20-minute pad test. Follow-up assessments will be conducted immediately after the fourth- and eighth-week treatment period and at a three-month post-treatment follow-up. During these assessments, participants will complete the same validated outcome measures as the baseline assessment to evaluate changes in genitourinary symptoms and quality of life following LLLT.

ELIGIBILITY:
Inclusion Criteria:

* Menopause women
* With genitourinary symptoms of menopause

Exclusion Criteria:

* Acute or chronic infection of the genitourinary tract
* Advanced pelvic organ prolapse (>= stage 2 on pelvic organ prolapse quantification system)
* History of pelvic malignancy
* Unstable blood pressure
* Fever
* Abnormal sensory nerve
* Abnormal coagulation

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal health | 20 weeks
  Vaginal health index, each of these 5 items is evaluated by means of a scale from 1 (none) to 5 (excellent) and then the average of the scores is calculated. A value of ≤15 (= cut-off) is generally considered for the diagnosis of low vaginal health.

SECONDARY OUTCOMES:
Lower urinary tract symptom: incontinence | 20 weeks
  ICIQ-SF: International Consultation on Incontinence Questionnaire - Short Form. Scoring scale: 0-21. Higher scores mean a worse outcome.
Lower urinary tract symptom: general | 20 weeks
  UDI-6: Urogenital Distress Inventory-6. Scoring scale: 0-18. Higher scores mean a worse outcome.
Lower urinary tract symptom: life quality | 20 weeks
  IIQ-7: Incontinence Impact Questionnaire-7. Scoring scale: 0-21. Higher scores mean a worse outcome.
Lower urinary tract symptom: urgency | 20 weeks
  USS: Urgency Severity Scale. The USS is scored as 0 (no feeling of urgency), 1 (mild urgency), 2 (moderate urgency), 3 (severe urgency), or 4 (inability to hold urine).
Lower urinary tract symptom: overactive bladder | 20 weeks
  OABSS: Overactive Bladder Symptom Score. The total score ranges from 0 to 15 points, with higher scores indicating higher symptom severity.
Quality of life affected by lower urinary tract symptoms | 20 weeks
  KHQ: King's Health Questionnaire. It addresses nine different domains in 21 items with a Likert scale response options (range 1-4 and 1-5 on the first option). The domains are general health perception, incontinence impact, role limitations, physical and social limitations, personal relationships, emotions, sleep/energy, and severity coping measures. An additional independent scale with nine questions was designed to evaluate symptom severity perception. Scores for each domain are calculated through a complex system that manages missing values and results range from 0 to 100, with higher scores indicating a more impaired QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-chi Wu, MD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The datasets analyzed during the study are available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: 3 years after finishing study.
Access Criteria: The datasets analyzed during the study are available from the PI upon reasonable request.

REFERENCES:
- [Background] Rola P, Doroszko A, Derkacz A. The Use of Low-Level Energy Laser Radiation in Basic and Clinical Research. Adv Clin Exp Med. 2014 September-October;23(5):835-842. doi: 10.17219/acem/37263. PMID 25491701
- [Result] Phillips NA, Bachmann GA. The genitourinary syndrome of menopause. Menopause. 2021 Feb 1;28(5):579-588. doi: 10.1097/GME.0000000000001728. PMID 33534428
- [Result] Gambacciani M, Palacios S. Laser therapy for the restoration of vaginal function. Maturitas. 2017 May;99:10-15. doi: 10.1016/j.maturitas.2017.01.012. Epub 2017 Feb 4. PMID 28364861
- [Result] Long CY, Wu PC, Chen HS, Lin KL, Loo Z, Liu Y, Wu CH. Changes in sexual function and vaginal topography using transperineal ultrasound after vaginal laser treatment for women with stress urinary incontinence. Sci Rep. 2022 Mar 2;12(1):3435. doi: 10.1038/s41598-022-06601-0. PMID 35236871
- [Result] Filippini M, Porcari I, Ruffolo AF, Casiraghi A, Farinelli M, Uccella S, Franchi M, Candiani M, Salvatore S. CO2-Laser therapy and Genitourinary Syndrome of Menopause: A Systematic Review and Meta-Analysis. J Sex Med. 2022 Mar;19(3):452-470. doi: 10.1016/j.jsxm.2021.12.010. Epub 2022 Jan 29. PMID 35101378
- [Result] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033